CLINICAL TRIAL: NCT05738707
Title: Clinical Study of SARS-CoV-2 Vaccine Sequentially Enhancing Immune Response in Metabolism-related Fatty Liver Disease Based on Deep Machine Learning
Brief Title: Clinical Study of SARS-CoV-2 Vaccine in Metabolism-related Fatty Liver Disease
Status: Not yet recruiting | Type: Observational
Sponsor: The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School (Other)
Responsible Party: Principal Investigator, Jie Li, Principal Investigator, The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Other Study IDs: 2023-128
Record Dates: First submitted 2023-01-28; First posted 2023-02-22 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Metabolic Associated Fatty Liver Disease
Keywords: SARS-CoV-2; vaccination; immune response

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Recombinant protein vaccine
  Interventions: Biological: Recombinant protein vaccine and adenovirus vector vaccine
- Adenovirus vector vaccine
  Interventions: Biological: Recombinant protein vaccine and adenovirus vector vaccine

INTERVENTIONS:
Biological: Recombinant protein vaccine and adenovirus vector vaccine — Administer recombinant protein vaccine and adenovirus vector vaccine

SUMMARY:
The coronavirus disease 2019 (COVID-19) caused by SARS-CoV-2 causes high morbidity and mortality worldwide. SARS-CoV-2 vaccination is currently the most effective means of reducing morbidity, severe illness and mortality risk. This study aimed to establish a metabolic associated fatty liver disease (MAFLD) cohort of sequential booster SARS-CoV-2 vaccination, and to identify the dynamic changes of immune response induced by sequential booster SARS-CoV-2 vaccination in MAFLD population. To investigate the effects of blood routine, liver function biochemistry and coagulation function at 28 days, 57 days and 180 days after inoculation of SARS-CoV-2 vaccination.

DETAILED DESCRIPTION:
The coronavirus disease 2019 (COVID-19) caused by SARS-CoV-2 causes high morbidity and mortality worldwide. SARS-CoV-2 vaccination is currently the most effective means of reducing morbidity, severe illness and mortality risk. Metabolic associated fatty liver disease (MAFLD) has a prevalence rate of 29.63% in China, which is the most common chronic liver disease in China. This study aimed to establish a metabolic associated fatty liver disease (MAFLD) cohort of sequential booster SARS-CoV-2 vaccination, and to identify the dynamic changes of immune response induced by sequential booster SARS-CoV-2 vaccination in MAFLD population. To investigate the effects of blood routine, liver function biochemistry and coagulation function at 28 days, 57 days and 180 days after inoculation of SARS-CoV-2 vaccination. Safety and adverse events were assessed using an electronic questionnaire at days 1, 3, 5, and 7 after enrollment. Serum and peripheral blood PBMC were collected at baseline and 28, 57, and 180 days after vaccination. Blood routine, liver function biochemistry, coagulation function, antibodies, peripheral blood cell subtypes and serum, and PBMC proteomics were tested to evaluate the antibody and immune response induced by SARS-CoV-2 vaccination.

ELIGIBILITY:
Inclusion Criteria:

1. Strengthened by the third dose of SARS-CoV-2 vaccination in MAFDL population.
2. Age ≥18 years old, gender unlimited.
3. Persons who agree to participate in this clinical trial and sign informed consent voluntarily.

Exclusion Criteria:

1. Persons who failed to complete SARS-CoV-2 vaccination.
2. Start vaccination but do not strictly follow the vaccination schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of 100 patients with MAFLD who had completed full inactivated vaccine for more than 6 months were given different sequential booster immunization regimens, including 50 patients receiving recombinant protein vaccine and 50 patients receiving adenovirus vector vaccine
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-02 (Estimated); Primary Completion 2026-01 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Dynamic monitoring of neutralizing antibody titers | 28 days
  Dynamic monitoring of neutralizing antibody titers induced by SARS-CoV-2 vaccination
Dynamic monitoring of neutralizing antibody titers | 57 days
  Dynamic monitoring of neutralizing antibody titers induced by SARS-CoV-2 vaccination
Dynamic monitoring of neutralizing antibody titers | 180 days
  Dynamic monitoring of neutralizing antibody titers induced by SARS-CoV-2 vaccination

SECONDARY OUTCOMES:
Dynamic monitoring of titers of antibodies (RBD, S1, S2 and ECD) | 28 days
  Dynamic monitoring of titers of antibodies (RBD, S1, S2 and ECD) against different spike protein antigens of SARS-CoV-2 vaccination
Dynamic monitoring of titers of antibodies (RBD, S1, S2 and ECD) | 57 days
  Dynamic monitoring of titers of antibodies (RBD, S1, S2 and ECD) against different spike protein antigens of SARS-CoV-2 vaccination
Dynamic monitoring of titers of antibodies (RBD, S1, S2 and ECD) | 180 days
  Dynamic monitoring of titers of antibodies (RBD, S1, S2 and ECD) against different spike protein antigens of SARS-CoV-2 vaccination

OTHER OUTCOMES:
Dynamic monitoring of CD4+ and CD8+T cell responses to S, N, M, and E proteins | 28 days
  Dynamic monitoring of CD4+ and CD8+T cell responses to S, N, M, and E proteins induced by SARS-CoV-2 vaccination
Dynamic monitoring of CD4+ and CD8+T cell responses to S, N, M, and E proteins | 57 days
  Dynamic monitoring of CD4+ and CD8+T cell responses to S, N, M, and E proteins induced by SARS-CoV-2 vaccination
Dynamic monitoring of CD4+ and CD8+T cell responses to S, N, M, and E proteins | 180 days
  Dynamic monitoring of CD4+ and CD8+T cell responses to S, N, M, and E proteins induced by SARS-CoV-2 vaccination